CLINICAL TRIAL: NCT02808403
Title: Long Term Post Marketing Specified Drug Use Result Survey for Evolocumab (AMG 145) in Japan
Brief Title: Long Term Post Marketing Specified Drug Use Result Survey for Evolocumab in Japan
Status: Completed | Type: Observational
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Other Study IDs: 20140409
Record Dates: First submitted 2016-06-07; First posted 2016-06-21 (Estimated); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Hypercholesterolemia; Familial Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia; Hyperlipoproteinemia Type II

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Evolocumab exposed: Patients for whom evolocumab is prescribed. Dosage, period (start/end date), frequency of injection (Every 2 weeks (Q2W), Every 4 weeks (Q4W)), drug withdrawal (Yes or No, date, reason) and injection site (upper arm, abdomen, thigh) of evolocumab will be collected.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention; observation of routine medical care

SUMMARY:
The purpose of this post-marketing survey is to obtain real-world information on the safety and effectiveness of evolocumab in Japan.

DETAILED DESCRIPTION:
The objectives of study are to 1) determine the incidence of adverse events and adverse drug reactions among patients receiving evolocumab for up to 2 years, and 2) identify and describe patient characteristics (e.g. demographics, medical history) associated with the safety and effectiveness of evolocumab therapy for the patients with Familial Hypercholesterolemia (Heterozygous or Homozygous) and Hypercholesterolemia in Japan

ELIGIBILITY:
Inclusion Criteria:

* Patients for whom evolocumab is prescribed at participating medical institutions in accordance with the approved Japan prescribing information (i.e., those with Familial Hypercholesterolemia (Heterozygous or Homozygous and Hypercholesterolemia who have high risk factors for cardiovascular event and do not respond sufficiently to HMGCoA reductase inhibitor (statin) for hypercholesterolemia).

Exclusion Criteria:

* No exclusion criteria are applied.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients for whom evolocumab is prescribed at participating medical institutions in accordance with the approved Japan prescribing information (i.e., those with Familial Hypercholesterolemia and Hypercholesterolemia who have high risk factors for cardiovascular event and do not respond sufficiently to Hydroxymethylglutaryl coenzyme A (HMG-CoA) reductase inhibitor (statin) for hypercholesterolemia.)
Sampling Method: Non-Probability Sample
Enrollment: 6000 (Actual)
Dates: Start 2016-06-24 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events and adverse drug reactions | 2 years
  The incidence of adverse events and drug reactions will be described using the same units (events per 1000 person-years). Adverse events (including seriousness and causal relations to drug or device), inclusive of reaction at local injection sites, and other safety information (e.g. overdose, lack of effectiveness, pregnancy and lactation with or without adverse event) will be described.
Laboratory values for LDL-C | 2 years
Laboratory values for HDL-C | 2 years
Laboratory values for total cholesterol | 2 years
Laboratory values for triglycerides | 2 years
Laboratory values for Apolipoprotein (Apo) A1 | 2 years
  This will be measured if feasible.
Laboratory values for Apolipoprotein (Apo) Apo B | 2 years
  This will be measured if feasible.
Laboratory values for Apolipoprotein (Apo) Apo E | 2 years
  This will be measured if feasible.
Laboratory values for lipoprotein(a) | 2 years
  This will be measured if feasible.

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (100):
- Japan (100):
  - Research Site, Ichinomiya, Aichi-ken
  - Research Site, Inuyama, Aichi-ken
  - Research Site, Kasugai, Aichi-ken
  - Research Site, Komaki, Aichi-ken
  - Research Site, Nagoya, Aichi-ken
  - Research Site, Tsushima, Aichi-ken
  - Research Site, Akita, Akita
  - Research Site, Yuzawa, Akita
  - Research Site, Asahi, Chiba
  - Research Site, Chiba, Chiba
  - Research Site, Chosei Gun, Chiba
  - Research Site, Ichihara, Chiba
  - Research Site, Ichikawa, Chiba
  - Research Site, Kisarazu, Chiba
  - Research Site, Matsudo, Chiba
  - Research Site, Matsuyama, Ehime
  - Research Site, Fukuoka, Fukuoka
  - Research Site, Itoshima, Fukuoka
  - Research Site, Kitakyushu, Fukuoka
  - Research Site, Omuta, Fukuoka
  - Research Site, Futaba Gun, Fukushima
  - Research Site, Iwaki, Fukushima
  - Research Site, Kōriyama, Fukushima
  - Research Site, Kani, Gifu
  - Research Site, Mino, Gifu
  - Research Site, Nagahama City, Gifu
  - Research Site, Fujioka, Gunma
  - Research Site, Kiryū, Gunma
  - Research Site, Takasaki, Gunma
  - Research Site, Fukuyama, Hiroshima
  - Research Site, Higashihiroshima, Hiroshima
  - Research Site, Hiroshima, Hiroshima
  - Research Site, Onomichi, Hiroshima
  - Research Site, Iwamizawa, Hokkaido
  - Research Site, Sapporo, Hokkaido
  - Research Site, Himeji, Hyogo Prefectural
  - Research Site, Kobe, Hyogo Prefectural
  - Research Site, Sanda, Hyogo Prefectural
  - Research Site, Kobe, Hyōgo
  - Research Site, Higashiibaraki Gun, Ibaraki
  - Research Site, Hitachi, Ibaraki
  - Research Site, Mito, Ibaraki
  - Research Site, Kahoku Gun, Ishikawa-ken
  - Research Site, Kanazawa, Ishikawa-ken
  - Research Site, Mukai-awagasaki, Ishikawa-ken
  - Research Site, Kitakami, Iwate
  - Research Site, Morioka, Iwate
  - Research Site, Kita Gun, Kagawa-ken
  - Research Site, Sakaidechō, Kagawa-ken
  - Research Site, Zentsujichó, Kagawa-ken
  - Research Site, Kagoshima, Kagoshima-ken
  - Research Site, Kanoya, Kagoshima-ken
  - Research Site, Fujisawa, Kanagawa
  - Research Site, Kawasaki, Kanagawa
  - Research Site, Miura, Kanagawa
  - Research Site, Yokohama, Kanagawa
  - Research Site, Yokosuka, Kanagawa
  - Research Site, Kumamoto, Kumamoto
  - Research Site, Yamaga, Kumamoto
  - Research Site, Kyoto, Kyoto
  - Research Site, Maizuru, Kyoto
  - Research Site, Uji, Kyoto
  - Research Site, Yosa Gun, Kyoto
  - Research Site, Ise, Mie-ken
  - Research Site, Tsu, Mie-ken
  - Research Site, Sendai, Miyagi
  - Research Site, Miyazaki, Miyazaki
  - Research Site, Matsumoto, Nagano
  - Research Site, Niigata, Niigata
  - Research Site, Ōita, Oita Prefecture
  - Research Site, Okayama, Okayama-ken
  - Research Site, Izumisano, Osaka
  - Research Site, Kawachi-Nagano, Osaka
  - Research Site, Osaka, Osaka
  - Research Site, Suita, Osaka
  - Research Site, Takaishi, Osaka
  - Research Site, Takatsuki, Osaka
  - Research Site, Saga, Saga-ken
  - Research Site, Taku, Saga-ken
  - Research Site, Ageo, Saitama
  - Research Site, Koshigaya, Saitama
  - Research Site, Saitama, Saitama
  - Research Site, Moriyama, Shiga
  - Research Site, Hamada, Shimane
  - Research Site, Nikkō, Tochigi
  - Research Site, Tokushima, Tokushima
  - Research Site, Chuoku, Tokyo
  - Research Site, Hachiōji, Tokyo
  - Research Site, Higashikurume, Tokyo
  - Research Site, Kodaira, Tokyo
  - Research Site, Ōta-ku, Tokyo
  - Research Site, Shibuyaku, Tokyo
  - Research Site, Shinagawa City, Tokyo
  - Research Site, Sinagawa Ku, Tokyo
  - Research Site, Taitoku, Tokyo
  - Research Site, Toshimaku, Tokyo
  - Research Site, Gobō, Wakayama
  - Research Site, Shingū, Wakayama
  - Research Site, Wakayama, Wakayama
  - Research Site, Kofu, Yamanashi

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the link below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- [Derived] Yokote K, Ako J, Kitagawa K, Osada N, Sheng F, Sonoda M, Teramoto T. Safety and Effectiveness of Low-Density Lipoprotein Cholesterol-Lowering Therapy With Evolocumab for Familial Hypercholesterolemia/Hypercholesterolemia in Japan: A Real-World, Postmarketing, Single-Arm Study. J Am Heart Assoc. 2024 Nov 5;13(21):e035809. doi: 10.1161/JAHA.124.035809. Epub 2024 Oct 29. PMID 39470058